CLINICAL TRIAL: NCT03700801
Title: Multicenter Prospective Cohort Study of the Hypoglycemic Efficacy, Weight Control, and Safety in Newly-diagnosed Type 2 Diabetes: Triple Combination Therapy Using Metformin, Saxagliptin Plus Dapagliflozin Versus Premixed Insulin
Brief Title: Study of Efficacy, Weight Control, and Safety in Newly-diagnosed Type 2 Diabetes With Different Antidiabetic Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Zhujiang Hospital (Other)
Collaborators: The Sixth Affiliated Hospital of Guangzhou Medical University (Other); Third Affiliated Hospital, Sun Yat-Sen University (Other); Peking University Shenzhen Hospital (Other); Dongguan Kanghua Hospital (Other); First People's Hospital, Shunde China (Other); The First Affiliated Hospital of Guangdong Pharmaceutical University (Other); The Fifth Affiliated Hospital of Zunyi Medical College (Other); Shenzhen Sixth People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-NFMDXK-003
Record Dates: First submitted 2018-09-09; First posted 2018-10-09 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2018-10

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Triple Combination Therapy; Premixed Insulin; Hypoglycemic efficacy; Weight control; Safety
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin; dapagliflozin; saxagliptin; insulin aspart, insulin aspart protamine drug combination 30:70

STUDY DESIGN:
Intervention Model Description: According to two different therapies, patients were divided into the study group (triple combination therapy group) and control group (premixed insulin treatment group). Each group included 65 cases.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Triple combination therapy group (Experimental): triple combination therapy group: Triple oral hypoglycemic therapy based on metformin 0.5mg twice a day, dapagliflozin 10mg per day plus saxagliptin 5mg per day.
  Interventions: Drug: Triple combination therapy group
- Premixed insulin therapy group (Active Comparator): premixed insulin therapy group: The initial total dose is 0.3U-0.5U/Kg, twice a day, subcutaneous injection before breakfast and dinner, adjusted according to the blood glucose level detected by the blood glucose meter
  Interventions: Drug: Premixed insulin therapy group

INTERVENTIONS:
Drug: Triple combination therapy group — Triple oral hypoglycemic therapy based on metformin, dapagliflozin plus saxagliptin.
  Other Names: Metformin, Dapagliflozin and Saxagliptin
  Arms: Triple combination therapy group
Drug: Premixed insulin therapy group — Subcutaneous injection therapy with insulin aspart 30 in patients with T2DM
  Other Names: Insulin aspart 30
  Arms: Premixed insulin therapy group

SUMMARY:
Study Hypothesis：Compared with premixed insulin, triple oral combination therapy has similar hypoglycemic effect, better weight control and lower incidence of hypoglycemia.

Main objective: Comparing whether the hypoglycemic efficacy of the triple oral combination therapy is not inferior than that of the premixed insulin in the treatment of newly-diagnosed type 2 diabetes.

Secondary objective: Comparing the effects on body weight and the risk of inducing hypoglycemia between triple oral combination therapy and premixed insulin, and exploring the effects of these two therapies on weight control and safety.

Primary Study Endpoint: The absolute change in baseline of HAb1c after 12 weeks.

Secondary Study Endpoint: fasting blood glucose, 2-hour postprandial blood glucose, fasting C-peptide, 2-hour postprandial C-peptide, body weight, proportion of patients with hypoglycemia, etc.

DETAILED DESCRIPTION:
Overview of research design：Newly diagnosed T2DM patients who meet the inclusion/exclusion criteria will be divided into a triple oral combination group (study group) or a premixed insulin treatment group (control group). Blood glucose of these two groups will be recorded during 12 weeks of treatment. And the change of the following effected indexes after 12 weeks of treatment will be recorded: HbA1c, fasting / 2-hour postprandial c-peptide. Also, weight, times of hypoglycemia and the occurrence of adverse events will be recorded during the whole study.

Details during implementation:

1. Grouping：

   In the cohort study, patients are divided into two groups, with the study group as the triple drug group and the control group as the premixed insulin treatment group. The grouping method is as follows:

   Non-randomized grouping method was performed in this study. After signing the informed consent, the participants were assigned a corresponding number according to the order in which they were included in the study. For example, if the patient was the first to be included in the cohort, his number was taken as No. 1; if the patient was the second to be included in the cohort, his number was taken as No. 2, and so on. Then patients were assigned to corresponding group based on their assigned numbers. If the assigned numbers were odd, they were arranged in triple combination therapy group; if not, they were arranged in premixed Insulin group.
2. Drugs treatment and dose adjustment:

   The use of saxagliptin: the initial dose is 5mg / time,1 time/day, before breakfast; if the blood glucose dose not reach the standard when metformin and dapagliflozin have been used up to the above-mentioned maximum amount, then adjust the dose in the order of "7.5mg / time, 1 time/day, taken before morning;10mg / time, 1 time/day, taken before breakfast" every 2 weeks; If the patient's blood glucose still fails to reach the standard with the initial dose of the above-mentioned triple combination in 2 weeks, the drug is adjusted to the maximum dose in the order of "metformin-daglipide-saxagliptin". If the blood glucose still fails to reach the standard, it is recommended that the patients quit the study and then switch to other hypoglycemic therapy; if hypoglycemia occurs during the incremental adjustment of the drug, and the effects of insufficient diet and excessive exercise are excluded, it is recommended to maintain the therapeutic dose before the dose of drug increased. If the patient has symptoms of hypoglycemia (dizziness, fatigue, hand tremor, palpitations, etc.) when taking the initial dose of the above-mentioned triple drug, it is considering to be the result of insufficient eating or excessive exercise, then patients need temporarily eating to correct hypoglycemia and investigators emphasize again to the patient the education in diet, sports, etc. If the patient's diet is normal and the factors of excessive exercise are excluded, adjust the drug treatment plan by firstly halving the dose of dapagliflozin, and closely monitor the patient's blood glucose for the next week: if the blood glucose does not reach the standard, continue to use the original triple therapy (metformin 0.5g/time 2 times/day or 3 times/day + saxagliptin 5 mg/time 1 time/day + dapagliflozin 10 mg/time 1 time/day); if the blood glucose reaches the standard and no hypoglycemia symptoms occurs, maintain the existing plan (Metformin 0.5g / time 2 times/day or 3 times/day + saxagliptin 5mg/time 1 time/day + dapagliflozin 5mg/time 1 time/day), and monitor blood glucose every week for not less than 2 days; If hypoglycemia still occurs, the dose of saxagliptin should be reduced by half (metformin 0.5g /time 2 /day or 3 /day + saxagliptin 2.5mg/time 1 /day + dapagliflozin 5mg/time 1 /day). If hypoglycemia still occurs, reduce the dose of metformin to 0.5g /time 1 /day. If hypoglycemia still occurs, then the patient will withdraw from the test, the medication is used according to the actual situation of the patient and the patient's glucose is continue to be monitored to ensure the glucose level of the patient reach the standard smoothly.

   Insulin aspart 30: The initial total dose is 0.3U-0.5U/Kg, 2 times/day, subcutaneous injection before breakfast and dinner, adjusted according to the blood glucose level detected by the blood glucose meter. The target of insulin aspart 30 is that fasting fingertip blood glucose (FBG) <7mmol/L, postprandial fingertip blood glucose (PBG) <10mmol/L after three meals, if the blood glucose still not reach the standard (the blood glucose measured in the specified monitoring time is not within the above range two days in a row), then the clinical physicians adjust the insulin treatment therapy based on the patient's blood glucose level, including increasing or decreasing the dose of insulin aspart 30.

   During the above-mentioned premixed insulin treatment, if hypoglycemia symptoms (dizziness, fatigue, hand tremor, palpitations, etc.) occur caused by insufficient eating or excessive exercise, then patients need temporarily eating to correct hypoglycemia and investigators emphasize the diet and sport again to the patient. If the patient's diet is normal and the factors of excessive exercise are excluded, then the premixed insulin dose is lowered by 2-4 IU/time.
3. Blood glucose monitoring:

   The patient prepares the blood glucose meter and test paper at home, and the researchers will explain to them how to use the device and give them adequate training. Self-monitoring of blood glucose will be carried out by patients themselves at home. The frequency of blood glucose monitoring is set as follows: monitoring frequency is once a day for the first week; twice a day for the second week; once every three days for the third and fourth weeks. After that, if blood glucose reaches the standard and remains stable, it is recommended for patients to monitor blood glucose at least one day a week; If blood glucose can't reach the standard or is unstable, the frequency of monitoring is at least once every three days for recommendation.

   Glycemic control standard refers to fasting fingertip blood glucose (FBG) <7mmol/L and postprandial fingertip blood glucose (PBG) <10mmol/L, without presenting of hypoglycemia (blood sugar <3mmol/L) and associated symptoms (dizziness, fatigue, tremor, palpitations, etc.) Detection time for fingertip blood glucose: fasting, 2 hours after breakfast, before bedtime.

   During each telephone follow-up, the researcher will record the patient's blood glucose, adverse events, and guide the patient to handle hypoglycemia, such as measure the blood glucose, eat cookies and candy rapidly, and record them in a log, whenever hypoglycemia symptoms appear
4. Follow-up At lease four times of visit：The first visit would last relatively longer with around 4 days to screen and confirm appropriate volunteers. And the next three visits, four weeks a day are mainly to assess the health for subjects. Additionally, subjects are required to have a HbA1c test in the first and last visit.

Telephone follow-up: During the study period, the investigators will conduct a weekly telephone follow-up of the subjects to find out their medication records, blood glucose levels and adverse events, and to adjust their medication dosage in time in case of adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. The newly-diagnosed type 2 diabetes mellitus according to the 1999 WHO guideline on diagnosing type 2 diabetes mellitus; 9%≤HbA1c≤12%;
2. Age: 18-65 years old, Men or women;
3. Voluntarily taking the triple combination therapy using metformin, saxagliptin plus dapagliflozin or premixed insulin therapy, without taking any other hypoglycemic therapy before;
4. 18.5kg/m2≦BMI≦32 kg/m2;
5. Voluntarily participating in our study and insisting on monitoring blood glucose at least one day a week, finishing re-examination after three month with the informed consent signed.

Exclusion Criteria:

1. Type 1 diabetes mellitus, or islet dysfunction (fasting C-peptide <0.1nmol/L (0.3ng/ml), peak value <0.17nmol/L (0.5ng/ml))
2. Patients with acute complication：ketoacidosis / hyperglycemic hyperosmolar status / lactic acidosis.
3. Patients with proliferative diabetic retinopathy.
4. Patients with severe infection or urinary tract infection.
5. Patients with clinically significant hepatobiliary disorders, including but not limited to chronic active hepatitis and / or severe liver dysfunction. ALT or AST> 3 times the normal upper limit (ULN) or serum total bilirubin (TB)> 34.2 μmol / L (> 2 mg / dL).
6. Patients with the following nephrotic history or kidney disease-related characteristics：

   1. history of unstable or acute kidney disease;
   2. Patients with moderate / severe renal injury or end-stage renal disease (eGFR <60 mL / min / 1.73 m2)
   3. urinary albumin: creatinine ratio> 1800 mg / g;
   4. the serum (Cr) ≥133 μmol / L (≥1.50 mg / dL) in male subjects; the serum Cr≥124μmol / L (> 1.40 mg / dL) in female subjects;
   5. congenital renal glucosuria;
7. Poor control of Severe hypertension, SBP ≥ 160 mmHg and / or DBP ≥ 100 mmHg; SBP <96 mmHg;
8. Patients with myocardial infarction / unstable angina / severe arrhythmia / heart failure in the past 3 months;
9. Hb≤110g/L in female subjects and Hb≤120g/L in male subjects;
10. Pregnant women or women who are planning to be pregnant during the study, women who are currently in lactation, or who having not adopted highly effective, medical-approved birth control methods.
11. Gastrointestinal diseases or surgical history, including Roemheld syndrome, severe hernia, intestinal obstruction, intestinal ulcers, gastrointestinal anastomosis, bowel resection, weight loss surgery or banding surgery;
12. Taking any drugs that affect blood sugar or body weight, history of alcohol or drug abuse over the past 6 months;
13. Patients who have received organ transplants or who have been definitely diagnosed as immunodeficiency syndrome with immune disfunction;
14. With a history of hypersensitivity or contraindication to metformin, saxagliptin, dapagliflozin or other drugs to be used in the researched.
15. Patients that might not follow this program, or with severe physical/mental illness that may affect the effectiveness or safety, based on the judgement of investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
HbA1c | 12 weeks
  Changes in HbA1c after 12 weeks of intervention.

SECONDARY OUTCOMES:
fasting/2-hour postprandial blood glucose | 12 weeks
  Changes in fasting/2-hour postprandial blood glucose after 12 weeks of intervention.
Fasting/2-hour postprandial c-peptide | 12 weeks
  Changes in fasting/2-hour postprandial c-peptide after 12 weeks of intervention.
Weight | 12 weeks
  Change in weight after 12 weeks of intervention.
Rate of hypoglycemia | 12 weeks
  Rate of hypoglycemia in two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Jia Sun, Study Director — Department of Endocrinology, Zhujiang Hospital, Southern Medical University
Locations (1):
- The Pearl River Hospital of Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No